CLINICAL TRIAL: NCT02348151
Title: Analysis of Metabolic and Ventilatory Demands During the Shuttle Walk Test Performed on a Treadmill Versus a Corridor in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Shuttle Walk Test Performed on a Treadmill Versus a Corridor in Patients With COPD
Acronym: (SWTiCOPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Patricia Lira dos Santos, Patricia Lira dos Santos, University of Nove de Julho
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: DPOCPC
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; SWTi; Treadmill
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treadmill (Experimental): The Shuttle is going to play on treadmill
  Interventions: Other: Treadmill
- Corridor (Active Comparator): The Shuttle is going to play on corridor
  Interventions: Other: Corridor

INTERVENTIONS:
Other: Treadmill — The volunteers will perform the shuttle walk test on the treadmill
  Arms: Treadmill
Other: Corridor — The volunteers will perform the shuttle walk test on the corridor
  Arms: Corridor

SUMMARY:
It is still not clearly known whether doing the walk test in a course is different from doing it on a treadmill in the lack of a ten-meter-long corridor. In case of a positive outcome in this study, we will have an alternative for this test in places where there is not enough room, benefiting the assessment of COPD patients' functional capacity. In the literature, there are still some controversies about performing the test on a treadmill or in a corridor and whether there is interference with the distance walked. Our hypothesis is that there is no interference with the distance walked, and thus we have one more option to perform the test in case there is no 10-meter corridor available.

DETAILED DESCRIPTION:
Spirometry tests will be performed using ULTIMA CPX equipment. Volunteers will perform the tests twice, on different days (see protocol description), in a corridor and on a treadmill, until reaching their limit of tolerance. In the test performed on the treadmill and in the one performed in the corridor, subjects will simultaneously use the VO 2000. And the volunteers will fill out the Saint George's Respiratory Questionnaire (SGRQ).

ELIGIBILITY:
Inclusion Criteria:

* clinically stable
* not dependent on oxygen to exercise
* diagnosis of COPD according to the GOLD

Exclusion Criteria:

* cognitive deficit or musculoskeletal
* in process of exacerbation
* have performed pulmonary rehabilitation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The distance reached in shuttle walk test | two year

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia L Santos, Professional, Principal Investigator — 551198408-4006
Locations (1):
- Patricia Lira dos Santos, Mogi das Cruzes, São Paulo/Mogi Das Cruzes, Brazil

REFERENCES:
- [Result] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Result] Stevens D, Elpern E, Sharma K, Szidon P, Ankin M, Kesten S. Comparison of hallway and treadmill six-minute walk tests. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1540-3. doi: 10.1164/ajrccm.160.5.9808139. PMID 10556117